CLINICAL TRIAL: NCT01607151
Title: Safety and Feasibility of a Protocol of Targeted Temperature Management After Intracerebral Hemorrhage
Brief Title: Safety and Feasibility Study of Targeted Temperature Management After ICH
Acronym: TTM-ICH
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thomas Jefferson University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12CRP12050342
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Intracerebral Hemorrhage
Keywords: hypothermia; normothermia; hyperthermia
MeSH Terms: conditions — Cerebral Hemorrhage; Hypothermia; Hyperthermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normothermia (Active Comparator): Core temperature 36-37 C
  Interventions: Other: Normothermia
- Hypothermia (Experimental): Core temperature 32-34 C
  Interventions: Other: Hypothermia

INTERVENTIONS:
Other: Normothermia — 72 hours of targeted temperature management to achieve normothermia (36-37°C)
  Arms: Normothermia
Other: Hypothermia — 72 hours of targeted temperature management to achieve hypothermia (32-34°C)
  Arms: Hypothermia

SUMMARY:
Though TTM is ubiquitously used in the neuro-intensive care unit, there is limited experience with the use of TTM after intracerebral hemorrhage (ICH), the most devastating type of stroke. TTM may be a an intervention to improve patient outcomes. This trial addresses the safety and tolerability of a protocol of ultra-early TTM after ICH/IPH and may be the basis for future larger clinical trials.

DETAILED DESCRIPTION:
Morbidity and mortality from intra-cerebral/intra-parenchymal hemorrhage (ICH/IPH) are important public health problems. As the most common etiology of ICH/IPH is hypertension, this places a large proportion of the population at risk. In 2011 The American Heart Association (AHA) estimated that in the US, there were 610,000 new stroke cases of which 10% were ICHs, and many required long-term health care. ICH/IPH is associated with the highest morbidity and mortality and only 20% of patients regain functional independence. Temperature modulation to hypothermia (T, 32-34°C) has been associated with modulation of physiopathologic processes associated with inflammatory activation and degradation of blood-brain barrier after all types of brain injury. Currently, there are no therapies to specifically target ICH/IPH. To this end, novel strategies that go beyond control of glucose, blood pressure, and intra-cranial pressure, aimed at reducing the enlargement of the hematoma and "swelling" surrounding it, could be "the new frontier in the management of ICH/IPH". Since the early resuscitation phase in the Neuro-ICU represents the greatest opportunity for impact on clinical outcome after ICH/IPH, it also appears to be the most promising window of opportunity to demonstrate a benefit when investigating novel therapies.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous supratentorial ICH documented by CT scan within 18 hours after the onset of symptoms
* Admission to the Neuro-ICU
* Baseline hematoma >15cc with or without IVH
* Need for mechanical ventilation.

Exclusion Criteria:

* GCS <6
* Age <18 years
* Pregnancy
* Pre-morbid modified Rankin Scale (mRS) >2
* Do Not Resuscitate (DNR) order "prior" to enrollment
* Uncontrolled bleeding of different etiology (trauma, gastro-intestinal bleeding [UGIB/LGIB])
* Planned surgical decompression within 24 hours
* Secondary causes of ICH (ischemic stroke, coagulopathy [INR>1.4, aPTT> 1.5 times baseline, thrombocytopenia platelets <100,000/uL], trauma, AVM, aneurysm, cerebral sinus thrombosis, or other causes)
* Evidence of sepsis
* Spontaneous hypothermia (core Temperature <36C)
* Inability to obtain written informed consent
* Participation in another trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Severe adverse events (SAEs) | 90 days
  The primary outcome measures will be: a) the frequency of adverse events (AEs) that will be possibly or probably related to treatment. AEs will be assessed up to 15-days after admission or discharge if earlier, and b) the frequency of severe adverse events (SAEs) that will be possibly and probably related to treatment.

SECONDARY OUTCOMES:
In-hospital neurological deterioration between day 0-7 | 7 days
  Decrease in GCS in ≥2 points or increase in the NIHSS ≥4 points
Functional outcome | Discharge and 90 days
  Modified Rankin Scale at discharge and 90-days.
Hematoma growth | 24 hours
  Absolute change in hematoma between baseline and 24 hours CT-scan and new or absolute change in IVH between baseline and 24 hours CT-scan
Cerebral edema | 24, 48,72, and 168-hours
  The absolute change in cerebral edema and the relative change in cerebral edema (absolute edema/absolute ICH volume unit less ratio)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Rincon, MD, MSc, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States